CLINICAL TRIAL: NCT04671862
Title: Photobiomodulation for the Prevention of Oral Mucositis in Patients Treated With Radiotherapy for Head and Neck Cancer
Brief Title: Photobiomodulation for the Prevention of Radiation Induced Oral Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190729-01H
Record Dates: First submitted 2020-11-18; First posted 2020-12-17 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Mucositis Oral; Head and Neck Cancer; Radiation Dermatitis
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Radiodermatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photobiomodulation (Experimental): Parameters: combined 633nm and 870 nm @1000mW
  * 1 Treatment pre radiotherapy
  * 3 treatments weekly during radiotherapy
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Parameters: combined 633nm and 870 nm @1000mW
  * 1 Treatment 4J continuous prior to RT. (Within 14 days of RT start)
  * 3 treatments weekly during RT (6 J at 12 Hz, 80% duty cycle)

SUMMARY:
Radiotherapy for head and neck cancer can cause severe mucositis (ulcers in the mouth) and pain. Photobiomodulation (Light therapy) will be used before and during radiotherapy to try to reduce the occurence and severity of mucositis in patients treated with radiotherapy for head and neck cancer

Previous studies in head and neck cancer patients have shown that photobiomodulation (light therapy) can prevent mucositis. There are currently no centers in Canada using this technique in routine practice, but this is recommended in International guidelines and widely used in Europe. The investigators therefore wish to implement this technique in Ottawa under the umbrella of a clinical trial to insure its safety and efficacy in a Canadian context.

DETAILED DESCRIPTION:
Introduction: Radiotherapy for head and neck cancer can cause severe mucositis (ulcers in the mouth) and pain. Photobiomodulation (Light therapy) will be used before and during radiotherapy to try to reduce the occurence and severity of mucositis in patients treated with radiotherapy for head and neck cancer

Rationale: Previous studies in head and neck cancer patients have shown that photobiomodulation (light therapy) can prevent mucositis. There are currently no centers in Canada using this technique in routine practice, but this is recommended in International guidelines and widely used in Europe. The investigators therefore wish to implement this technique in Ottawa under the umbrella of a clinical trial to insure its safety and efficacy in a Canadian context.

Purpose/Objectives: Primary Objective Primary Objective

• To determine the cumulative incidence of acute mucositis as defined by CTCAE version 2.0 for radiation induced mucositis (Appendix 1) during radiotherapy and for 1month following radiotherapy

Secondary Objectives

To determine the following during radiotherapy and for 24 months post-treatment

* Rate of occurrence of acute radiation dermatitis
* Pain scores
* Opioid use
* ESAS scores during and after RT
* FACT-HN questionnaire scores
* Late subcutaneous neck fibrosis
* Late mucosal and skin telangiectasia

Study design/methodology:

This is single arm prospective cohort study of a single intervention (photobiomodulation) in patients with head and neck cancer for the prevention of oral mucositis.

Outcomes will be the following:

* Rates of acute and late mucositis according to CTCAE version 2.0
* Rates of acute and late dermatitis and fibrosis according to CTCAE version 5.0
* Rates of late teleangiectasia
* Pain scores as per Edmonton Symptom assessment scale (ESAS) and modified brief pain inventory
* Rates of opioid use
* FACT-HN scores
* EQ5D scores

Anticipated public/scientific benefit:

This study aims to study the use of Photobiomodulation treatments for prevention of oral mucositis. This is recommended in international guidelines but not used in routine practice in Canada. The benefit of this study is to allow implemetation of this technique in the Canadian context in a controlled and evaluated manner. This will hopefully then allow further study and wider implementation of this technique both in Ottawa and in Canada

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Willing and able to understand and sign informed consent form approved by the institutional review board (IRB)
* Histological diagnosis of head and neck cancer of the oral cavity with no evidence of macroscopic residual disease post-surgery (R0 or R1 resection) and no gross residual lymphadenopathy in the planned PBM treatment area
* Planned treatment with radiotherapy or chemoradiotherapy to a dose of ≥ 50 Gy
* ECOG Performance Status of 0 or 1
* Intact oral mucosa (no visible ulceration, dehiscence or active infection

Exclusion Criteria:

* Gross macroscopic residual disease post surgery (R2 resection) or gross residual lymphadenopathy in the planned PBM treatment area
* Prior radiotherapy to the Head and Neck including the oral or oropharyngeal mucosa.
* Prior cytotoxic chemotherapy in the last 3 months
* Diagnosis of photosensitive disorder (cutaneous porphyria, xeroderma pigmentosum, etc)
* Concurrent administration of Cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of occurence of radiation mucositis | 7-14 days post radiotherapy
  CTCAE version 2.0
Rate of occurence of radiation mucositis | 1 month post radiotherapy
  CTCAE version 2.0
Rate of occurence of radiation mucositis | 3 months post radiotherapy
  CTCAE version 2.0
Rate of occurence of radiation mucositis | 6 months post radiotherapy
  CTCAE version 2.0
Rate of occurence of radiation mucositis | 12 months post radiotherapy
  CTCAE version 2.0
Rate of occurence of radiation mucositis | 24 months post radiotherapy
  CTCAE version 2.0

SECONDARY OUTCOMES:
Brief Pain Inventory | 7-14 days post radiotherapy
  Pain questionnaire
Brief Pain Inventory | 1 month post radiotherapy
  Pain questionnaire
Brief Pain Inventory | 3 months post radiotherapy
  Pain questionnaire
Brief Pain Inventory | 6 months post radiotherapy
  Pain questionnaire
Brief Pain Inventory | 12 months post radiotherapy
  Pain questionnaire
Brief Pain Inventory | 24 months post radiotherapy
  Pain questionnaire
Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) | 7-14 days post-radiotherapy
  Swallowing related quality of life
Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) | 1 month post-radiotherapy
  Swallowing related quality of life
Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) | 3 months post-radiotherapy
  Swallowing related quality of life
Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) | 12 months post-radiotherapy
  Swallowing related quality of life
Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) | 24 months post-radiotherapy
  Swallowing related quality of life
EQ-5D | 7-14 days post radiotherapy
  General Quality of life questionnaire
EQ-5D | 1 month post radiotherapy
  General Quality of life questionnaire
EQ-5D | 3 months post radiotherapy
  General Quality of life questionnaire
EQ-5D | 6 months post radiotherapy
  General Quality of life questionnaire
EQ-5D | 12 months post radiotherapy
  General Quality of life questionnaire
EQ-5D | 24 months post radiotherapy
  General Quality of life questionnaire
Radiation dermatitis | 7-14 days post radiotherapy
  CTCAE version 5.0
Radiation dermatitis | 1 month post radiotherapy
  CTCAE version 5.0
Radiation dermatitis | 3 months post radiotherapy
  CTCAE version 5.0
Radiation dermatitis | 6 months post radiotherapy
  CTCAE version 5.0
Radiation dermatitis | 12 months post radiotherapy
  CTCAE version 5.0
Radiation dermatitis | 24 months post radiotherapy
  CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No